CLINICAL TRIAL: NCT04308356
Title: "What if we Talked About it…" Identification of Cancer Patients Taking up a Proposal for Discussions Dedicated to Anticipating Preferences of Care in the Event of Aggravation (DDA): Prospective Cohort Intervention Study Using a Mixed Methodology
Brief Title: Do Patients Want to Engage in Discussions Dedicated to Anticipating (DDA) Their Preferences of Care in the Event of Worsening Health Status?
Acronym: ESOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190416; 2019-A01802-55 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-06; First posted 2020-03-16 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Neoplasm Metastasis; Locoregional Neoplasm; Advanced Cancer
Keywords: Prospective monocentric cohort study; Mixed methodology; Dedicated Discussions on Anticipating preferences; Care; Aggravation
MeSH Terms: conditions — Neoplasm Metastasis | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Dedicated Discussions on Anticipating preferences of care in the event of Aggravation (DDA) — interview 2
Other: Autonomy Preference Index (API ) questionnaire - Information — part of interview 1
Other: anxiety and depression (HADS) questionnaire — part of interview 1

SUMMARY:
Context: In people concerned by serious illness, how to anticipate the aggravation of the disease according to the patient's preferences is a challenging clinical question and an ethical key-issue to improve end-of-life care and quality of dying in France. When end of life decision occurs, many patients can no longer express themselves and advance directives do not seem to be appropriate for many patients despite the current strong incentives to write them, reinforced by the 2016 Claeys Leonetti.

The "End-of-Life Discussions" and "Advance care planning" programs developed in the United States have shown a positive impact on the aggressiveness of end-of-life care. The implementation in France of these programs has not yet been consolidated despite a first recommendation for "Planification des soins futurs", published by the French Health Authority(HAS). Inspired by the definition given in the later document, investigators propose the acronym DDA, for the Discussions Dedicated to Anticipate wishes and preferences in the event of Aggravation, defined as the dynamic and evolving process of reflection and communication between the patient, his relatives and healthcare professionals, allowing him to address his preferences and wishes regarding his care and treatment

The objective of this observational study is to characterize, in a population of patients with advanced cancer, the profile of those who take up a proposal for Dedicated Discussions on Anticipating preferences of care in the event of Aggravation (DDA) and who engage in the discussion process. Secondary objectives are to

1. evaluate the aggressiveness of end-of-life care in the group of patients who died 1 year after their inclusion, depending on their engagement in DDA occurs and whether or not their preferences are formalized; and
2. evaluate the subjective effects of the DDA with the patient and the investigating professionals, through qualitative approach by a clinical psychologist.

Method: investigators designed a mixed, quantitative and qualitative prospective, monocenter methodology to evaluate how patients take up a proposal of DDA. This proposal consists in 2 interviews: the first one is dedicated to the assessment of the patient's wishes in terms of information and participation in decision-making (API questionnaire) and to the assessment of the degree of anxiety and depression (HADS questionnaire) (E1). The second one is conducted 1 to 4 weeks later and consists in offering and initiating DDA (E2).

Quantitative outcome evaluated will be:

1. the documentation by a physician in the medical record, of patient's care preferences/values
2. the documentation by the patient of his care preference/values, either by designation of surrogate or by writing advanced directives
3. the usefulness and necessity of this approach, and the anxiety it generated, as perceived by the patient The qualitative assessment will be based on data collected during E1 and E2, and for 20 patients, during a clinical interview with a psychologist dedicated to collecting the patient's impressions of previous interviews.

Thanks to this study investigators expect to gather some data on the desire and feelings of cancer patients to engage in a DDA process and possibly formalize their end-of-life preferences, the impact of DDAs on care pathway indicators and the psychological effect for the patient with severe disease to project himself in advance into aggravation.

These expected results will provide a better understanding of the process of anticipating end-of-life situations, which is needed to improve quality of care and end-of-life conditions.

DETAILED DESCRIPTION:
In the United States, the respect of patient's autonomy was early considered in 1990 by the Patient Self Determination Act, which stated that all persons entering a publicly funded health care facility had to be informed of their rights to formulate living wills. Meanwhile, tools have been developed to evaluate patients' expectations regarding information and participation in medical decision-making, e.g. the Autonomy Preference Index (API), initially conceived for general practice [Ende J 1989]. Since then, "End-of-Life Discussions" and "Advance care planning" programs have shown a positive impact on the aggressiveness of end-of-life care [Wright 2008, Mack 2012, Dow 2009]. However, some other studies have also suggested that patients in situations of real worsening would be less likely to seek prognostic information and could be unsettled by these programs [Michael 2013; Maciejewski 2013].

In France, the right to designate a "durable power of attorney for health care" (fr. "Personne de Confiance" (PC)) dates back to 2002, and the right to formulate "living wills" (fr. "Directives Anticipées" (DA)) concerning end-of-life care was first introduced by law in 2005 and their importance was reinforced in 2016. Recently, investigators established the validity and reliability of the French version of the API among patients with incurable cancer and in primary care setting. They found high patient expectations for information on their health status but a more variable desire to be involved in medical decisions. Three supplementary items were added specifically to evaluate incurable cancer patients' attitude towards anticipating their preference of care in the event of worsening health status. These suggested that anticipating may be for patients a specific dimension, not correlated with those of information and participation in decision making. Other French surveys show the low appropriation of PC and DA and suggest that DAs are not necessarily appropriate for all patients, despite the strong current incentives to write them.

The implementation in France of "Advance care planning" programs has not yet been consolidated despite a first recommendation for "Planification des soins futurs", published by the HAS (French Health Authority). Inspired by the definition given in the later document, we propose the acronym DDA, for the Discussions Dedicated to Anticipate wishes and preferences in the event of Aggravation, defined as the dynamic and evolving process of reflection and communication between the patient, his relatives and healthcare professionals, allowing him to address his preferences and wishes regarding his care and treatment.

Considering that the strictly numerical objective of writing living wills or designating a PC is not a relevant indicator of quality of care, investigators rather aim to get a better understanding of the process of DDA, assuming that this process would contribute to improve quality of care at the end-of-life.

The objective of this observational study is to characterize, in a population of patients with advanced cancer, the profile of those who take up a proposal for Dedicated Discussions on Anticipating preferences of care in the event of Aggravation (DDA) and who engage in the discussion process. Secondary objectives are to 1) evaluate the aggressiveness of end-of-life care in the group of patients who died 1 year after their inclusion, depending on their engagement in DDA occurs and whether or not their preferences are formalized; and 2) evaluate the subjective effects of the DDA with the patient and the investigating professionals, through qualitative approach by a clinical psychologist.

For each of 240 patients with advanced metastatic cancer recruited in the oncology department of a university hospital, the mixed method of evaluation consists in :

* collecting their preferences thanks to the API, along with their degree of anxiety/depression (HADS scale) (interview E1)
* initiating DDA (interview E2)
* collecting their evaluation of E2 by quantitative criteria (self-reported anxiety, perceived usefulness,…) and their qualitative subjective impressions on E1 and E2 (by clinical psychologist in a subgroup of 20 patients)
* following up their engagement in the DDA process and its impact on healthcare resource use in the last month of life (quantitative outcomes).

Quantitative outcomes evaluated were inspired by the results of the consensus work published by Sudore and al, on outcomes design to evaluate success of Advance Care Planning. There will be:

1. the documentation by a physician in the medical record, of patient's care preferences/values
2. the documentation by the patient of his care preference/values, either by designation of surrogate or by writing advanced directives
3. the usefulness and necessity of this approach, and the anxiety it generated, as perceived by the patient The qualitative assessment will be based on data collected during E1 and E2, and for 20 patients, during a clinical interview with a psychologist dedicated to collecting the patient's impressions of previous interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Followed by oncologists from the medical oncology and pulmonology departments of Cochin Hospital,
* with advanced stage cancer (solid neoplasm, any location) (locoregional or metastatic),
* whose objective of care is not curative (in the sense of healing)
* whose life expectancy is less than 1 year, estimated by the investigating physician, by the standard question, commonly used in the literature, "would you be surprised if this patient died within the next year?"

Exclusion Criteria:

* Severe psychopathology (generalized anxiety disorder, panic disorder, schizophrenia spectrum disorders, bipolar and related disorders, and major depressive disorders), mentioned in the patient medical record
* Persistent cognitive disorders, with type of dementia or confusion, mentioned in the patient medical record
* Patient not fluent in French
* Eastern Cooperative Oncology Group (ECOG) Performance status = 4
* A refusal of the patient after proposal and information about the study
* Patient not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients population in medical care for advance cancer in oncology or pneumology, for which the aim is not the cure of the disease, but rather longer survival or quality of life maintenance, whose lifespan expectation is approximately higher than a year.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Documentation by a physician of patient's care preferences/values 6 months after E2 interview | 7 months
  Rate of patients for whom this documentation by a physician is found in hospital electronic medical record

SECONDARY OUTCOMES:
Patient has decided and documented his/her choice on a surrogate decision maker | 7 months
  Rate of patients who have designated their surrogate on the appropriate form, signed by both the patient and surrogate
Patient has written advanced directives | 7 months
  Rate of patients who either declare having written advanced directives at E2 OR at telephone interview 2 months after E2 OR for whom advances directives are documented in their hospital electronic medical record 6 months after E2
Patient has discussed values and care preferences with the surrogate | 7 months
  Rate of patients who declare having discussed this with their surrogate, as investigated at the E2 interview
Anxiety generated by the E2 interview | at the end of E2 (4 weeks)
  Patient-reported anxiety, on a numerical scale (0 no anxiety-10 maximal imaginable anxiety)
REASSURING | at the end of E2 (4 weeks)
  answer "YES" to the question: "Do you think this interview and discussion was REASSURING?
NECESSITY | at the end of E2 (4 weeks)
  answer "YES" to the question: "Do you think this interview and discussion was NECESSARY?
USEFULNESS | at the end of E2 (4 weeks)
  answer "YES" to the question: "Do you think this interview and discussion was USEFUL?
Complete initiation of DDA | at the end of E2 (4 weeks)
  Rate of patients who completed the E2 interview until its end (with all data specified collected)
Time from 1st intervention of the palliative care team to death <30 days | 12 months follow-up
  Evaluated only in decedents (i.e early access to palliative care)
Proportion of patients who received chemotherapy in the last 14 days of life | 12 months follow-up
  Evaluated only in decedents
Proportion of patients who visited ≥2 times emergency room in the last month of life | 12 months follow-up
  Evaluated only in decedents
Proportion of patients admitted at least once to intensive care in the last month | 12 months follow-up
  Evaluated only in decedents
Time from transfer to Palliative Care Inpatient Unit (if applicable) to death <= 3 days | 12 months follow-up
  Evaluated only in decedents, (i.e. late transfer to Palliative Care Inpatient Unit)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle COLOMBET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Unité Fonctionnelle de Médecine palliative, Hôpitaux Universitaire Paris Centre - CHU Cochin, Paris, France

REFERENCES:
- [Background] Sudore RL, Heyland DK, Lum HD, Rietjens JAC, Korfage IJ, Ritchie CS, Hanson LC, Meier DE, Pantilat SZ, Lorenz K, Howard M, Green MJ, Simon JE, Feuz MA, You JJ. Outcomes That Define Successful Advance Care Planning: A Delphi Panel Consensus. J Pain Symptom Manage. 2018 Feb;55(2):245-255.e8. doi: 10.1016/j.jpainsymman.2017.08.025. Epub 2017 Sep 1. PMID 28865870
- [Background] Michael N, O'Callaghan C, Clayton J, Pollard A, Stepanov N, Spruyt O, Michael M, Ball D. Understanding how cancer patients actualise, relinquish, and reject advance care planning: implications for practice. Support Care Cancer. 2013 Aug;21(8):2195-205. doi: 10.1007/s00520-013-1779-6. Epub 2013 Mar 14. PMID 23494583
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Mack JW, Cronin A, Keating NL, Taback N, Huskamp HA, Malin JL, Earle CC, Weeks JC. Associations between end-of-life discussion characteristics and care received near death: a prospective cohort study. J Clin Oncol. 2012 Dec 10;30(35):4387-95. doi: 10.1200/JCO.2012.43.6055. Epub 2012 Nov 13. PMID 23150700
- [Background] Dow LA, Matsuyama RK, Ramakrishnan V, Kuhn L, Lamont EB, Lyckholm L, Smith TJ. Paradoxes in advance care planning: the complex relationship of oncology patients, their physicians, and advance medical directives. J Clin Oncol. 2010 Jan 10;28(2):299-304. doi: 10.1200/JCO.2009.24.6397. Epub 2009 Nov 23. PMID 19933909
- [Background] Maciejewski PK, Prigerson HG. Emotional numbness modifies the effect of end-of-life discussions on end-of-life care. J Pain Symptom Manage. 2013 May;45(5):841-7. doi: 10.1016/j.jpainsymman.2012.04.003. Epub 2012 Aug 25. PMID 22926093